CLINICAL TRIAL: NCT06434415
Title: Prognostic Value of Coronary Angiography-Derived Index of Microcirculatory Resistance in Hypertrophic Cardiomyopathy Patients
Brief Title: Prognostic Value of Angio-IMR in Hypertrophic Cardiomyopathy Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024005
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-05

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCM patients with low angio-IMR: This group patients have low angio-IMR value in LAD.
- HCM patients with high angio-IMR: This group patients have high angio-IMR value in LAD.

SUMMARY:
Coronary microvascular dysfunction (CMD) is among pathophysiological states of significance in hypertrophic cardiomyopathy (HCM). The index of microcirculatory resistance (IMR) has been recognized as an indicator of CMD and considered of important prognostic value in various conditions. The angiography-derived index of microcirculatory resistance (angio-IMR) is a novel guidewire-free method to assess IMR and proved to have favourable correlation with it. This study was designed to assess prognostic impact of CMD in HCM patients, using angio-IMR as a novel non-invasive assessment tool.

DETAILED DESCRIPTION:
Coronary microvascular dysfunction (CMD) is among pathophysiological states of significance in hypertrophic cardiomyopathy (HCM). The index of microcirculatory resistance (IMR) has been recognized as an indicator of CMD and considered of important prognostic value in various conditions. The angiography-derived index of microcirculatory resistance (angio-IMR) is a novel guidewire-free method to assess IMR and proved to have favourable correlation with it. In this study, patients who met the inclusion criteria were collected from two centers, and the angio-IMR of three coronary arteries was measured to monitor their microcirculation. Then, explore the prognostic value of the angio-IMR of the left anterior descending artery (LAD). At the same time combined with the sum of three coronary arteries' angio-IMR, analysis of its prognostic value. In conclusion, this study was designed to assess prognostic impact of CMD in HCM patients, using angio-IMR as a novel non-invasive assessment tool.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with hypertrophic cardiomyopathy(HCM) based on clinical guidelines
2. have qualified image for analysis of angio-IMR

Exclusion Criteria:

1）referred to hospital due to ST-segment elevation myocardial infarction(STEMI), heart failure and cardiopulmonary arrest; 2) Implantation of any DES or DCB; 3）severe valve dysfunction; 4）history of implantation of implantable cardioverter-defibrillator or pacemaker, septal myectomy or septal myocardial ablation; 5）meet the criteria of implantation of implantable cardioverter-defibrillator or pacemaker, septal myectomy or septal myocardial ablation; 6）impaired life-span expectancy due to cancer or other clinical conditions；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively enrolled patients who were diagnosed with hypertrophic cardiomyopathy(HCM) and underwent invasive coronary angiography between 2017 and 2024 at two sites (The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China; Ningbo Medical Center Lihuili Hospital, Ningbo, China) .The diagnosis of HCM was based on current clinical guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
MACE composite | within 24 months' follow-up
  a composition of death from cardiovascular causes, progression to severe functional limitation (NYHA class III or IV), and sustained, life-threatening ventricular arrhythmias requiring the implantation of a cardioverter-defibrillator,septal myocardial ablation or septal myectomy, new on stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jiang, MD, PhD, Study Director — Second affiliated Hospital Zhejiang University School of Medicine